CLINICAL TRIAL: NCT02866045
Title: Endoscopic Ultrasonography Guided Fine Needle Biopsy (EUS-FNB) vs. Single-incision Needle-knife (SINK) Biopsy for Diagnosis of Upper Gastrointestinal Subepithelial Lesions
Brief Title: EUS-FNB vs. Single-incision Needle-knife (SINK) Biopsy for Gastrointestinal SELs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 16-030
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Disorder of Upper Gastrointestinal Tract; Gastrointestinal Stromal Tumors; Gastrointestinal Neoplasms
Keywords: Subepithelial lesions; Endoscopic Ultrasound-Guided Fine Needle Aspiration
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-guided Fine Needle Biopsy (Active Comparator): EUS-FNB is performed using a 22 or 25 G SharkCore biopsy needle with a minimum of 3 passes into the lesion.
  Interventions: Procedure: EUS-guided fine needle biopsy
- Single incision needle knife biopsy (Experimental): SINK biopsy is performed under direct endoscopic visualization via EGD with a minimum of 3 biopsy samples obtained.
  Interventions: Procedure: Single incision needle knife biopsy

INTERVENTIONS:
Procedure: EUS-guided fine needle biopsy — EUS-FNB is performed using a 22 or 25 G core biopsy needle (SharkCore FNB, Medtronic, Fridley, MN) by standard linear EUS-guided technique. The needle tip has six cutting edge surfaces and an opposing bevel to catch tissue as it is sheared off, enabling cohesive units of tissue acquisition with minimal tissue fracturing. 3 separate passes will be done into the lesion. Additional passes may be made if clinically necessary. No suction will be applied on the first pass. If the FNB sample obtained is deemed to be inadequate, negative pressure (using the standard suction syringe) will be applied to the needle on additional passes. The histology and cytology specimens will be processed as per standard clinical care.
  Other Names: EUS-FNB
  Arms: EUS-guided Fine Needle Biopsy
Procedure: Single incision needle knife biopsy — For patients allocated to the SINK group, after EUS confirmation, the esophagogastroduodenoscopy (EGD) will be repeated to perform the SINK biopsy. Under direct endoscopic visualization, a 10 mm linear incision will be made to the surface of the SEL using a conventional needle-knife sphincterotome with standard blended electrocautery (Endocut mode - ERBE system USA, Marietta, GA). A conventional biopsy forceps will then be introduced through the incision deep into the mass to obtain at least 3 samples. The incision will then be closed using 1 to 3 endoclips for prophylaxis against subsequent bleeding. The biopsies will be placed in formalin as per standard surgical pathology protocol.
  Other Names: SINK
  Arms: Single incision needle knife biopsy

SUMMARY:
Sub epithelial lesions (SELs) of the gastrointestinal (GI) tract are commonly identified during routine endoscopy. Most of these lesions are benign. However because there is the potential for malignant transformation it is important to correctly identify the lesion in order to determine if any further therapy and/or surveillance is necessary for the patient, particularly for gastrointestinal stromal tumors (GISTs).

Obtaining a definitive diagnosis for SELs is often difficult since biopsies of the normal overlying surface mucosal layer are typically normal. EUS-FNA is the standard method by which a biopsy-proven diagnosis is obtained for most SEL's. However, the yield for a definite diagnosis from EUS-FNA for SELs is often suboptimal. Recently a new biopsy method, called "single incision needle-knife" (SINK) was introduced that may prove more useful in determining a definitive diagnosis. Furthermore, recent advances in core biopsy needles for EUS offer the hope for improved outcomes with EUS-guided fine-needle biopsy (FNB). However, it remains unclear whether superior diagnostic outcomes are obtained using the new SINK biopsy method or using new EUS-FNB core needles.

DETAILED DESCRIPTION:
Subepithelial lesions of the gastrointestinal (GI) tract are commonly identified during routine endoscopy. Most of these lesions are benign. However because there is the potential for malignant transformation it is important to correctly identify the lesion in order to determine if any further therapy and/or surveillance is necessary for the patient.

Leiomyoma, neural origin tumors, lipoma, duplication cyst, pancreatic rest, inflammatory fibroid polyp, granular cell tumor are considered benign SELs. Gastrointestinal stromal tumor, lymphoma, carcinoid, metastatic carcinoma, glomus tumor are malignant or potentially malignant lesions. Obtaining a diagnosis for SELs is often difficult since biopsies of the normal overlying surface mucosal layer are typically normal. Jumbo forceps biopsy, bite-on-bite technique with conventional biopsy forceps, endoscopic ultrasound (EUS) guided fine needle aspiration (FNA), fine needle biopsy (FNB), single incision needle-knife biopsy (SINK), and endoscopic resection allow sampling of deeper tissue layers and may provide a histologic diagnosis. However there are no standard biopsy methods to diagnose SELs.

Endoscopic ultrasound (EUS) is a helpful imaging diagnostic tool for the evaluation of SELs as it is capable of assessing its size, layer of origin, and echo patterns. However, it is not reliable enough to differentiate between benign and malignant SELs. The combination of EUS and fine needle aspiration (FNA) allows for cytologic diagnostic accuracy of about 80%. If a malignant tumor is suspected, tissue acquisition is important because the management may vary based on the type of SEL.

EUS-FNA enables a small needle to be passed into the lesion of interest under ultrasound guidance, obtaining cellular material for cytology analysis. Although previous reports show accuracy rates for EUS-FNA for SEL that range between 72% and 90% there often is a problem of inadequate cellular aspirates for additional immunocytochemical examination. This problem causes a miss rate of approximately 40% for additional immunocytochemical analyses that may be needed to reach a definitive diagnosis for GISTs, although the macroscopic appearance alone is often sufficient. Using a larger FNA needle to perform the biopsy seems to be a logical solution to this limitation. However, doing so has thus far not been shown to improve the adequacy of biopsy aspirates.

For this reason, core biopsy needles (EUS-FNB) have been developed in the hopes of obtaining core tissue for histology. The advantages of a biopsy core specimen are well known because the evaluation of tissue architecture increase the diagnostic yield compared to cytology obtained from FNA. In addition, a tissue core biopsy is critical to diagnose and characterize SELs by providing higher rates of immunohistological evaluation. Recently, a novel design core biopsy needle (Sharkcore, Medtronic) has been introduced with preliminary data suggesting superior diagnostic performance compared to previous versions of core biopsy needles. How this new needle performs in the diagnostic evaluation of SELs remains unclear.

Single-incision needle-knife (SINK) biopsy is an alternative diagnostic method to acquire tissue samples. By using a conventional needle knife sphincterotome, the overlying mucosa of SELs is opened with a single linear incision of 10 mm and tissue samples are obtained by passing conventional biopsy forceps through the opening and deep into the tumor. According to a preliminary study by de la Serna Higuera et al, this technique provides sufficient tissue samples with high diagnostic yield of 92.8%. However, this biopsy method is only possible when a visible bulge from the SEL is apparent within the lumen of the gastrointestinal tract.

The investigators believe this technique offers the potential to obtain more substantial tissue samples that will be much more likely to provide a definitive diagnosis for subepithelial tumors. In addition, it is hoped that biopsy samples obtained via SINK will be better able to provide adequate tissue for determination of the mitotic rate of GIST tumors, which is a major predictor of malignant risk for these lesions. However, how the SINK method compares to the latest EUS-FNB core needles is unclear, both in terms of the diagnostic efficacy in obtaining the diagnosis and in terms of the safety profile of doing so.

The purpose of this study is to prospectively compare the efficacy and safety of EUS-FNB using the new SharkCore needle with SINK biopsy in patients with upper GI SELs. The results of the study will determine which method should be performed to confirm the diagnosis for SELs.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing diagnostic endoscopy for gastrointestinal SELs
* Tumor size ≥ 15 mm with endoscopically visible bulge
* SELs in esophagus, stomach, or duodenum
* Ability to sign the informed consent for diagnostic procedure

Exclusion Criteria:

* Lesions not requiring pathological evaluation (e.g. lipoma, cyst, varices)
* Underlying medical condition that contraindicates diagnostic endoscopy.
* Bleeding diathesis
* Inability to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving a definitive histologic diagnosis for gastrointestinal SELs by single incision needle-knife biopsy (SINK biopsy) vs. EUS-guided fine needle biopsy (EUS-FNB). | 24 months
  Percentage of patients in each group for whom the pathologist provides a definite histologic diagnosis based on the biopsy sample.

SECONDARY OUTCOMES:
Adverse events with SINK biopsy vs. EUS-FNB | 24 months
Procedure time with SINK biopsy vs. EUS-FNB | 24 months
Proportion of patients receiving a definite OR suspicious diagnosis for gastrointestinal SELs using SINK biopsy vs. EUS-FNB | 24 months
  Percentage of patients in each group for whom the pathologist provides a "definite" or "suspicious" histologic diagnosis based on the biopsy specimen.
Proportion of patients for whom a mitotic rate may be calculated for gastrointestinal stromal tumors (GISTs) using SINK biopsy vs. EUS-FNB | 24 months
  Percentage of patients in each group with a diagnosis of GIST for whom a mitotic rate may be calculated by the pathologist from the biopsy specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Teshima, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de la Serna-Higuera C, Perez-Miranda M, Diez-Redondo P, Gil-Simon P, Herranz T, Perez-Martin E, Ochoa C, Caro-Paton A. EUS-guided single-incision needle-knife biopsy: description and results of a new method for tissue sampling of subepithelial GI tumors (with video). Gastrointest Endosc. 2011 Sep;74(3):672-6. doi: 10.1016/j.gie.2011.05.042. PMID 21872716
- [Background] Mekky MA, Yamao K, Sawaki A, Mizuno N, Hara K, Nafeh MA, Osman AM, Koshikawa T, Yatabe Y, Bhatia V. Diagnostic utility of EUS-guided FNA in patients with gastric submucosal tumors. Gastrointest Endosc. 2010 May;71(6):913-9. doi: 10.1016/j.gie.2009.11.044. Epub 2010 Mar 11. PMID 20226456